CLINICAL TRIAL: NCT07361055
Title: The Best Workflow for Paroxysmal Supraventricular Tachycardia Ablation With Zero-fluoroscopy
Acronym: zeroPSVT
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Johnson & Johnson (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202401199RIPB
Record Dates: First submitted 2026-01-06; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-03

CONDITIONS: Cardio Vascular Disease; Cryoablation
Keywords: zero-fluoroscopy; paroxysmal supraventricular tachycardia ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Protocol A (Fam DX+) (Experimental): Create geometry FAM Mapping with DECANAV(Fam DX+)
  Interventions: Device: Protocol A
- Protocol B (FAM DX-) (Active Comparator): Create geometry FAM MAPPING WITH NAVISTAR (FAM DX-)
  Interventions: Device: Protocol B

INTERVENTIONS:
Device: Protocol A — Mapping with DECANAV
  Other Names: FAM DX+; DECANAV®
  Arms: Protocol A (Fam DX+)
Device: Protocol B — Mapping with NAVISTAR
  Other Names: FAM DX-; NAVISTAR®
  Arms: Protocol B (FAM DX-)

SUMMARY:
Primary Objective: To observe, record, and analyze the workflow and guidance system efficiency of these two surgical procedures, including placement time, location, and the number of successful placements.

Secondary Objective: To compare the differences between the two procedures and observe and record the process of transitioning to intracardiac ultrasound guidance by experienced physicians performing both workflows. The primary focus is on the time spent on target steps and related complications, with the aim of reducing radiation exposure during the procedure with the new technology.

DETAILED DESCRIPTION:
The aim of this study is to compare the safety and efficiency of two workflows (with or without FAM Dx) using CARTO® 3 System for PSVT ablation. The results will later be compared with another 3-dimentional mapping system (Ensite™) historically

ELIGIBILITY:
Inclusion Criteria:

1. Patients with documented PSVT on ECG. Twelve-lead is preferred. Single-lead is acceptable if recording quality is good enough for interpretation.
2. Patients who are willing to sign the informed consent.

Exclusion Criteria:

1. The patients had received PSVT ablation procedure before.
2. Informed consent could not be obtained

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-03-26 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
The success of ablation | 1Year
  defined by elimination of accessory pathway and slow nodal pathway or modification of the slow nodal pathway with which a PSVT upto 3 reentrants would not be induced

SECONDARY OUTCOMES:
The complication rates | 1Year
  including the occurrence of AV block needing pacemaker, or pericardial effusion needing drainage, or use of fluoroscopy

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospita, Taipei, Taiwan